CLINICAL TRIAL: NCT00664950
Title: A Multi-centre Randomized Control Trail Comparing a Novel Intramedullary Device (InterTAN) Versus Conventional Treatment (Sliding Hip Screw) of Geriatric Fractures.
Brief Title: InterTAN IM Nail Versus Sliding Hip Screw in Geriatric Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Orthopaedic Research Foundation (Other)
Responsible Party: Principal Investigator, David Sanders, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-08-002; 13619 (Other: REB)
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Hip Fractures
Keywords: intertrochanteric hip fracture fixation; interTAN IM Nail; sliding hip screw
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SHS (Active Comparator): sliding hip screw
  Interventions: Device: sliding hip screw
- InterTAn IM Nail (Active Comparator): interTAN IM nail
  Interventions: Device: IntertAn IM nail

INTERVENTIONS:
Device: sliding hip screw — surgical repair of hip fracture using conventional sliding hip screw
  Arms: SHS
Device: IntertAn IM nail — interTAN IM nail
  Other Names: InterTAn
  Arms: InterTAn IM Nail

SUMMARY:
Elderly patients with an intertrochanteric hip fracture will be randomized to receive either a sliding hip screw (SHS) (control group) or InterTAN intermedullary nail (IMN) (experimental group) for surgical fixation of their hip fracture. This study will assess functional and mortality outcomes for elderly patients with hip fractures.

DETAILED DESCRIPTION:
Outcome after hip fracture in the elderly is generally poor. According to the World Health Organization, fracture of the hip is associated with 20 % 1-year mortality and 50 % loss of function33. However, the high mortality and loss of function can be improved. For example, numerous studies have shown improvement in relevant outcomes when interventions such as improved thromboprophylaxis, care pathways and timely surgery are achieved. Up to 50 % decreases in mortality can be achieved with these interventions1,2,3.

While improvements in perioperative care can improve outcome, the benefit of newer surgical techniques and implants is less clear. This is well demonstrated in the case of intertrochanteric fractures. Intertrochanteric fractures are those in which the primary fracture line occurs between the greater and lesser trochanter and include approximately 50 % of all hip fractures. Many surgical implants have been developed for this common fracture pattern; in general, the conventional implant is a sliding hip screw (SHS) in which a plate is fixed to the lateral cortex of the femur, distal to the fracture; and a large-diameter screw is placed in the centre of the femoral head, proximal to the fracture. The screw and plate slide relative to one another, permitting compression of the fracture and facilitating bone healing. In contrast, the newer implants are typically intramedullary nail designs (IMN), in which a metal nail is placed within the canal of the femur and a large-diameter screw is placed in the centre of the femoral head. The theoretical advantage of newer designs is based upon, first, an improved stability of the implant, allowing earlier and more aggressive mobilization; and second, a less invasive surgical procedure to minimize blood loss. Nonetheless, repeated trials and meta-analyses have failed to demonstrate an advantage to the IMN designs compared to SHS. In fact, perioperative complications seem to be higher using the IMN designs4,5.

There are two primary reasons why IMN designs have not translated into improved results to date. First, perioperative complications, especially fractures of the femur, are more common with current IMN designs. Second, the supposed improved stability conferred by these devices may not actually be achieved. Current IMN designs retain the original concept of a single screw in the femoral head, which does not prevent rotation of the femoral head - a common reason for implant failure. As well, most current IMN designs permit unrestricted axial shortening of the femur, which may lead to significant leg length changes and alter gait.

A new implant has been designed to take advantage of the inherent theoretical strengths of IMN designs and improve upon current design flaws. The InterTAN device (IT) has been designed to improve stability after fixation of intertrochanteric fractures. This device has a double proximal hip screw, to achieve rotational control; improved implant geometry, to improve immediate stability; and immediate compression to achieve stability while avoiding uncontrolled leg length changes. The IT device retains the percutaneous insertion technique of other IMN devices and simplifies insertion with redesigned instrumentation. The InterTAN device is the first device designed specifically to provide enhanced stability to intertrochanteric fractures and seems to offer significant promise compared to other IM designs.

The InterTAN device has not, as of yet, been compared to conventional surgical techniques. According to the Cochrane Database Reviews, "Any new design should be evaluated in a randomised comparison with the sliding hip screw."

ELIGIBILITY:
Inclusion Criteria:

1. Age 55 years or greater*
2. Intertrochanteric fracture amenable to treatment by sliding hip screw or intramedullary nail fixation
3. Previously ambulatory (defined as not usually requiring a wheelchair for ambulation)*
4. Provision of informed consent*
5. Surgery performed within 72 hours of admission

Exclusion Criteria:

1. Cognitive or language barriers that would limit completion of assessment tests in English*
2. Anticipated problems with follow-up in the judgment of the resident, or attending surgeon (e.g of no fixed address)*
3. Surgeon refusal to randomize patient
4. Pathologic fractures
5. Polytrauma that would impact functional assessments in the opinion of the surgeon

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-11; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | prospective
Timed up an go (TUG) | prospective

SECONDARY OUTCOMES:
2-minute walk test (2MWT) | prospective
Geriatric Depression Scale (GDS) | prospective
Lower Extremity Measure (LEM) | prospective
Complications | prospective
Femoral shortening | prospective
Blood Loss | prospective
Mortality | prospective

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Dianne Bryant, Principal Investigator — Western University, Canada
Locations (3):
- Canada (3):
  - Saint John Regional Hosptial, Saint John, New Brunswick
  - London Health Sciences Centre, London, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario